CLINICAL TRIAL: NCT06723717
Title: Efficacy of Daily IV Administration of Dornase Alfa Up to 14 Days Post Subarachnoid Hemorrhage on Functional Independence At 6 Months: a PROBE Multicenter Open-label Randomized Controlled Trial
Brief Title: Efficacy of Daily IV Administration of Dornase Alfa Up to 14 Days Post Subarachnoid Hemorrhage on Functional Independence At 6 Months
Acronym: RESET
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FDE-2023-11
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ruptured Aneurysm of Intracranial Artery; SAH (Subarachnoid Hemorrhage); Delayed Cerebral Ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dornase alfa (Experimental): Daily infusion of dornase alfa at a dose of 125 microg/kg as an IV bolus until day 14 after SAH, on top of usual care
  Interventions: Drug: Daily infusion of dornase alfa
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Drug: Daily infusion of dornase alfa — Daily infusion of dornase alfa at a dose of 125 microg/kg as an intravenous bolus until day 14 after SAH
  Arms: Dornase alfa

SUMMARY:
Subarachnoid hemorrhage due to aneurysm rupture (SAH) results in high mortality, while survivors frequently suffer reduced quality of life and even loss of autonomy, particularly in the active population. A significant proportion of this morbidity and mortality is linked to the occurrence of delayed cerebral ischemia (DCI), defined as a new focal neurological deficit or reduced level of consciousness unrelated to the treatment of the aneurysm or a concomitant condition.

DCI mainly occurs between days 4 and 14 after SAH, with an estimated incidence of 30%, and is significantly associated with an unfavorable functional prognosis at 3 months. Currently, the only treatment for post-SAH DCI is to prevent or reverse the onset of vasospasm, with limited efficacy, for example through nimodipine administration or hemodynamic optimization. However, according to existing data, vasospasm is not the only cause of DCI, as it may occur elsewhere than in the arterial territory affected by vasospasm, or even in the absence of any vasospasm at all. Recent reviews of the literature highlight the role of microvascular thrombo-inflammation in the pathophysiology of DCI.

This phenomenon begins as soon as SAH occurs, with the appearance of multiple microvascular obstructions responsible for ischemia of downstream territories and loss of distal autoregulatory capacity. Among the effectors of thrombo-inflammation, the NETose phenomenon (production of NETs - Neutrophil Extracellular Traps or extracellular DNA network) has recently been associated with the onset of DCI. Indeed, the concentration of NETs increases in the cerebrospinal fluid (CSF) and blood of SAH patients, and correlates with the severity of the hemorrhage. Furthermore, intravenous or intraperitoneal administration of DNAse in an animal model of SAH has been shown to reduce NET concentration and improve functional prognosis by acting directly on cerebral perfusion through the reduction of micro-thrombosis.

In humans, recombinant DNAse (dornase alfa, Pulmozyme®) has marketing authorization for inhaled administration in cystic fibrosis. The toxicology report accompanying the marketing authorization demonstrates the absence of serious side effects following administration of high IV doses of Pulmozyme® in monkeys and rats. Other studies evaluating IV administration of bovine DNAse at high doses report no complications.

In 1999, a study was published evaluating intravenous (IV) Pulmozyme® in lupus patients, reporting no serious adverse events (SAEs) among the 14 patients receiving the treatment. We are currently conducting a clinical trial of the same molecule in IV administration in patients treated with mechanical thrombectomy and IV thrombolysis for ischemic stroke (NCT04785066).

This study is the first randomized clinical trial to target NETs as effectors of the thrombo-inflammation responsible for post-HSA DCI.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for subarachnoid hemorrhage (SAH) due to aneurysm rupture
* Onset of SAH symptoms less than 48 hours old
* Aneurysm exclusion performed within the last 24 hours
* No complications during exclusion procedure, confirmed on post-procedure CT scan
* Fisher score > 1 on initial brain CT scan prior to exclusion (first scan performed during emergency management)

Exclusion Criteria:

* Unidentified date of aneurysm rupture / rebleeding
* Severe infections
* Patient with impaired renal function (GFR < 60ml/min/1.73m2 or serum creatinine >1.5 mg/dL)
* Immediate complications of neurosurgical intervention or embolization
* Known hypersensitivity to dornase alfa, Chinese hamster ovary cell products or product excipients.
* Previous disability (mRS>1 prior to SAH)
* Pregnant or breast-feeding women (negative urine pregnancy test for women aged 49 or under)
* Participation in another interventional drug or medical device clinical trial within the 30 days prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Excellent functionnal independance at 6 months | Month 6
  Score of 0 or 1 on the modified Rankin Scale (mRS) at 6 months. Assessment will be centralized and performed by telephone by a certified professional, blinded to the randomization arm.
  mRS ranges from 0 to 6, 0 beeing total functionnal independance and 6 beeing death.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Delvoye, MD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild